CLINICAL TRIAL: NCT00807898
Title: Health Care Decisions for Female Adolescents: The Role of Mothers and Daughters in Decision Making
Status: Completed | Type: Observational
Sponsor: University of Louisville (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Mimia Logsdon, Professor, University of Louisville
Other Study IDs: OICB080587; Merck33563
Record Dates: First submitted 2008-12-11; First posted 2008-12-12 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2011-01

CONDITIONS: Cervical Cancer
Keywords: Gardasil; HPV vaccine; decision making; mother; daughter
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
Preventing cervical cancer is a public health concern. Since 2006 a quadrivalent vaccine for young women nine to twenty six years of age has been available to protect against the human papillomavirus (HPV) and to prevent some types of cervical cancer (Gardasil). The vaccine is an important health promotion tool to address the widespread prevalence of HPV and cervical cancer, but not all eligible young women receive the vaccine. The vaccine is most effective when administered to young women before their sexual debut. When the vaccine is given to young women less than 18 years of age, parental permission is required. This permission is usually provided by the young woman's mother. Understanding predictors of a mother's decision for her minor daughter to receive the HPV vaccine will inform interventions that seek to increase the number of young women who receive the vaccine.

The study will focus on mothers and their adolescent daughters between 13-17 years of age. We hypothesize that the Expanded Theory of Planned Behavior will explain a mother's decision to choose the HPV vaccine for her daughter.

Research Questions include: 1)What TPB variables predict a mother's decision to choose HPV vaccine for her daughter? 2)What variables predict the strength of a daughter's influence on the mother's decision to choose HPV vaccine for her daughter? 3) What are the relationships between the mothers' and daughters' scores on the variables related to the decision to choose HPV vaccine? 4) How do the mothers and daughters who chose to receive the HPV vaccine differ descriptively from those mothers and daughters who do not choose to receive the HPV vaccine?

DETAILED DESCRIPTION:
Preventing cervical cancer is a public health concern. Since 2006 a quadrivalent vaccine for young women nine to twenty six years of age has been available to protect against the human papillomavirus (HPV) and to prevent some types of cervical cancer (Gardasil). The vaccine is an important health promotion tool to address the widespread prevalence of HPV and cervical cancer, but not all eligible young women receive the vaccine. The vaccine is most effective when administered to young women before their sexual debut. When the vaccine is given to young women less than 18 years of age, parental permission is required. This permission is usually provided by the young woman's mother. Understanding predictors of a mother's decision for her minor daughter to receive the HPV vaccine will inform interventions that seek to increase the number of young women who receive the vaccine.

Health behavior theories, such as the Theory of Planned Behavior (TPB), indicate the factors and mechanisms that predict health promotion decisions and activities. TPB provides a direct statistical model through which variables related to health behaviors can be measured and evaluated, and will be used to guide the proposed study.

The study will focus on mothers and their adolescent daughters between 13-17 years of age. The normative changes and realignments in the parent child relationship that arrive with the onset of adolescence, coincide with greater adolescence behavioral autonomy, and influence over parental decisions related to the adolescent. Thus, we expanded the TPB to include the influence of the adolescent on the mother's decision for her daughter to receive the HPV vaccine.

Hypothesis: We hypothesize that the Expanded Theory of Planned Behavior will explain a mother's decision to choose the HPV vaccine for her daughter.

Research Questions:

RSQ1: What TPB variables predict a mother's decision to choose HPV vaccine for her daughter?

RSQ2: What variables predict the strength of a daughter's influence on the mother's decision to choose HPV vaccine for her daughter?

RSQ3: What are the relationships between the mothers' and daughters' scores on the variables related to the decision to choose HPV vaccine?

RSQ4: How do the mothers and daughters who chose to receive the HPV vaccine differ descriptively from those mothers and daughters who do not choose to receive the HPV vaccine?

Data will be analyzed using path analysis, multiple regression, and analysis of variance. The model demonstrates multiple potential influences on the mother's decision to choose the HPV vaccine for her daughter, and all influences are potential targets for family teaching interventions and tailored social marketing. Further study will be needed to determine how well the model applies to various family types and diverse cultures and nationalities.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent females 13-17 years of age
* and adolescent's mother, any age
* and adolescent not pregnant
* and adolescent has not received vaccine for HPV

Exclusion Criteria:

* Males
* daughters younger than 13 yrs of age
* daughters older than 17 yrs of age
* pregnant daughters
* daughters who have received the HPV vaccine

Min Age: 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Mother and daughter pairs (n =75) will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mimia C Logsdon, DNS, ARNP, FAAN, Principal Investigator — University of Louisville School of Nursing
Locations (1):
- University of Louisville School of Nursing, Louisville, Kentucky, United States

REFERENCES:
- [Derived] Hertweck SP, LaJoie AS, Pinto MD, Flamini L, Lynch T, Logsdon MC. Health care decision making by mothers for their adolescent daughters regarding the quadrivalent HPV vaccine. J Pediatr Adolesc Gynecol. 2013 Apr;26(2):96-101. doi: 10.1016/j.jpag.2012.10.009. PMID 23518189